CLINICAL TRIAL: NCT02609477
Title: A Double-Blind, Randomized, Placebo- and Active-Controlled Crossover Study to Evaluate the Abuse Potential of Istradefylline in Recreational Drug Users
Brief Title: A Study to Evaluate Abuse Potential of Istradefylline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 6002-017
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2016-08

CONDITIONS: Drug Abuse
Keywords: Recreational stimulant users; Recreational Drug Users
MeSH Terms: conditions — Substance-Related Disorders | interventions — istradefylline; Phentermine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Istradefylline 40 mg (Experimental): 40 mg istradefylline (1 × 40 mg tablet + 3 × placebo tablets + 3 × placebo capsules)
  Interventions: Drug: Istradefylline; Other: Placebo
- Istradefylline 80 mg (Experimental): 80 mg istradefylline (2 × 40 mg tablets + 2 × placebo tablets + 3 × placebo capsules)
  Interventions: Drug: Istradefylline; Other: Placebo
- Istradefylline 160 mg (Experimental): 160 mg istradefylline (4 × 40 mg tablets + 3 × placebo capsules)
  Interventions: Drug: Istradefylline; Other: Placebo
- Phentermine 45 mg (Active Comparator): 45 mg phentermine (4 x placebo tablets + 3 × 15 mg phentermine hydrochloride capsules)
  Interventions: Drug: Phentermine 45 mg; Other: Placebo
- Phentermine 90 mg (Active Comparator): 90 mg phentermine (4 × placebo tablets + 3 × 30 mg phentermine hydrochloride capsules)
  Interventions: Drug: Phentermine 45 mg; Other: Placebo
- Placebo (Placebo Comparator): Placebo (4 × placebo tablets + 3 × placebo capsules)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Istradefylline — Istradefylline 40, 80, 160 mg
  Other Names: 6002
  Arms: Istradefylline 160 mg; Istradefylline 40 mg; Istradefylline 80 mg
Drug: Phentermine 45 mg — Phentermine 45 or 90 mg
  Arms: Phentermine 45 mg; Phentermine 90 mg
Other: Placebo — Placebo

SUMMARY:
This study is to evaluate the abuse potential of single-doses of istradefylline compared to placebo and phentermine in recreational stimulant users. Subjects will participate in an outpatient medical Screening visit, a 5-day Qualification (Drug Discrimination) Phase, a 6-period Treatment Phase, and an outpatient safety Follow-Up visit. Study will be approximately 25 weeks total.

Within 28 days of the Screening visit, eligible subjects will be admitted to the CRU (Day -1) for the Qualification Phase. During the Qualification Phase, subjects will receive single oral doses of phentermine 60 mg and matching placebo in a randomized, double blind, crossover manner, with each drug administration separated by approximately 48 hours (Day 1 and Day 3), to ensure that they can discriminate and show positive subjective effects of the active controls. Following evaluation of eligibility, subjects may be discharged (those who fail Qualification criteria) or remain in the CRU (those who pass criteria and are eligible) and then proceed directly to the Treatment Phase. The washout interval between last drug administration in the Qualification Phase and first drug administration in the Treatment Phase will be at least 96 hours (4 days).

Following confirmation of eligibility from the Qualification Phase, subjects will be randomized to one of 6 treatment sequences according to a 6x6 Williams square. Subjects will receive single oral doses of each of the 6 treatments in a randomized, double-blind, crossover manner, Istradefylline 40 mg, Istradefylline 80 mg, Istradefylline 160 mg, Phentermine 45 mg, Phentermine 90 mg, Placebo.

Each drug administration will be separated by at least 21 days. Serial pharmacodynamic evaluations will be conducted up to 24 hours after each study drug administration to confirm exposure to istradefylline.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who will provide written informed consent
* Healthy volunteer, male and female between 18 and 55 years of age, inclusive
* Subjects with a body mass index (BMI) within 18.0 to 33.0 kg/m2, inclusive
* Subjects who are recreational drug user

Exclusion Criteria:

* Subjects who have an alcohol or substance dependence within the 12 months
* Subjects who have ever been in treatment for substance use disorder
* Subjects who consume on average more than 5 servings of caffeinated beverages per day
* Subjects with a history of or presence of any clinically significant cardiovascular disease
* Subject with hyperthyroidism or glaucoma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Drug Liking VAS | 24 hours
  To evaluate the abuse potential of istradefylline compared to phentermine and placebo.

SECONDARY OUTCOMES:
C-SSRS (Columbia Suicide Severity Rating Scale) | 24 hours
  To evaluate the safety and tolerability of istradefylline.
Alerness/Drowsiness, Agitation/Relaxation VAS | 24 hours
  To evaluate the safety and tolerability of istradefylline.
Caffine Withdrawal/Symptom Questionnaire | 24 hours
  To evaluate the safety and tolerability of istradefylline.
Overall Drug Liking, Take Drug Again VAS | 24 hours
  To evaluate the safety and tolerability of istradefylline.
Drug Similarity VAS | 24 hours
  To evaluate the safety and tolerability of istradefylline.

CONTACTS AND LOCATIONS:
Overall Officials: Kyowa Hakko Kirin Pharma, Inc., Study Chair — Kyowa Hakko Kirin Pharma, Inc.
Locations (1):
- Pharmaceutical Research Associates, Inc, Salt Lake City, Utah, United States